CLINICAL TRIAL: NCT06141577
Title: A Randomized, Open-label, Multiple-dose Crossover Phase 1 Clinical Trial to Compare and Evaluate the Safety, Pharmacokinetics and Pharmacodynamics Characteristics After Oral Administration of UI059 and UIC202201 in Healthy Adult Volunteers
Brief Title: A Study to Compare Pharmacokinetics, Pharmacodynamics and Safety of UI059 and UIC202201 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UI059-101
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, multiple-dose crossover phase 1 clinical
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UI059 (Experimental)
  Interventions: Drug: UI059
- UIC202201 (Active Comparator)
  Interventions: Drug: UIC202201

INTERVENTIONS:
Drug: UI059 — take UI059 1cap/day for 7 days
  Other Names: Test
  Arms: UI059
Drug: UIC202201 — take UIC202201 1cap/day for 7 days
  Other Names: Reference
  Arms: UIC202201

SUMMARY:
A randomized, open-label, multiple-dose crossover phase 1 clinical trial to compare and evaluate the safety, pharmacokinetics and pharmacodynamics characteristics after oral administration of UI059 and UIC202201 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers aged 19 and above.
* For males, a weight of 50.0 kg or more, and for females, a weight of 45.0 kg or more, with a body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2.

BMI(kg/m2)=Weight(kg)/height(m)2

* No congenital or chronic diseases requiring treatment, and no pathological symptoms or findings based on internal medicine examination.
* Those who were determined to be suitable subjects for clinical trials as a result of tests such as clinical laboratory tests, vital signs, physical examination (physical examination), and 12-lead electrocardiogram
* Negative for H. pylori antibodies
* After receiving detailed explanations about the clinical trial and fully understanding, participants voluntarily decide to participate and provide written consent to adhere to the subject compliance requirements throughout the trial period.

Exclusion Criteria:

* Current or past medical history of clinically significant conditions involving the liver, kidneys, nervous system, mental health, respiratory system, endocrine system, blood disorders, tumors, genitourinary system, cardiovascular system, digestive system, musculoskeletal system, etc., and in addition:

  * currently receiving antiretroviral drugs (rilpivirine, atazanavir, nelfinavir)
  * liver disorders
  * kidney disorders
* History of gastrointestinal conditions (Crohn's disease, ulcers, acute or chronic pancreatitis) or gastrointestinal surgery (excluding simple appendectomy or hernia repair) that may affect the absorption of the investigational drug.
* Pregnant (positive Urine-HCG) or lactating for female participants
* Have a history of hypersensitivity reactions (such as anaphylaxis or angioedema) or clinically significant hypersensitivity reactions to drugs, excipients, or other substances, including medications containing the active ingredients of the investigational drug, additives, and other drugs (such as aspirin, penicillin antibiotics, macrolide antibiotics).
* Have clinically significant findings on the 12-lead electrocardiogram during screening, including:

  * QTc interval > 450 ms for males or > 470 ms for females.
  * PR interval > 200 ms.
  * QRS duration > 120 ms.
* Showing the following results in clinical trial laboratory tests during screening:

  * liver function assessment: AST, ALT, ALP, γ-GTP, and total bilirubin exceeding twice the upper limit of the normal range.
  * Blood creatinine levels outside the reference range or calculated estimated glomerular filtration rate (eGFR) using the CKD-EPI formula less than 60 mL/min/1.73m2.
* History of drug abuse or individuals who have shown a positive reaction for abused substances in a urine drug test.
* During screening, exhibit vital signs measured after at least 3 minutes of rest in a seated position with systolic blood pressure (SBP) ≥ 150 mmHg or ≤ 90 mmHg, diastolic blood pressure (DBP) ≥ 100 mmHg or ≤ 60 mmHg, or a heart rate (HR) ≤ 40 bpm or ≥ 100 bpm.
* Have an abnormal diet that could affect the absorption, distribution, metabolism, or excretion of the investigational drug, or individuals who consume foods that could impact drug metabolism.
* Administered any prescription medications or herbal products that could influence the characteristics of the investigational drug within 2 weeks before the first dose or any OTC drugs or vitamin supplements within 10 days before the first dose. (If there is no effect on the pharmacokinetic properties of this investigational drug, the investigator may participate in the clinical trial at the discretion of the investigator.)
* Administer drugs that induce or inhibit drug-metabolizing enzymes, such as barbiturates, within 1 month before the first administration date.
* Participated in other clinical trials within 6 months prior to the first administration date (The endpoint for determining the end of participation in another clinical trial is considered one day after the last administration in that trial.)
* Those who have consistently consumed alcohol in excess of 21 units/week (1 unit = 10 g = 12.5 mL of pure alcohol) within 6 months prior to the first administration date or who are unable to abstain from alcohol from the time of written consent to the time of PSV.
* Smokers who smoke more than 10 cigarettes on average per day within 3 months before the first administration date and those who are unable to quit smoking from 24 hours before each administration until the time of the last blood collection
* Consumed food containing grapefruit or cannot refrain from eating it from 48 hours before the first administration until the time of PSV
* Those who consumed caffeine-containing foods (coffee, green tea, black tea, carbonated drinks, coffee milk, tonic drinks, etc.) during the period from 24 hours before administration to the time of the last blood collection, or who cannot refrain from consuming them.
* Those who engaged in vigorous exercise exceeding the level of daily life during the period from 48 hours before the first administration to the time of PSV, or who cannot refrain from vigorous exercise
* From the time of the subject's written consent until 2 weeks after the last administration of the investigational drug, even if the person, spouse, or partner is planning to become pregnant or is not planning to become pregnant, a recognized method of contraception (e.g., administration of contraceptives, implantation or intrauterine device, sterilization procedure (vasectomy), not using surgical resection, tubal ligation, etc.) or blocking methods (combined use of spermicides, condoms, contraceptive diaphragms, vaginal sponges, or cervical caps)
* Judged by the investigator to be unsuitable for participation in clinical trials due to reasons other than the above selection/exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss | Day 1: 0~24hours / Day 5, 6: 0hours / Day 7: 0~24hours
  Area under the plasma concentration-time curve within a dosing interval at steady state
Percent decrease from baseline in integrated gastric acidity | Day -1~Day 1, Day 1~Day 2, Day 7
  Percent decrease from baseline in integrated gastric acidity for 24 hours after multiple(7th dose) administrations

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Park, Dr, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk national university hospital, Cheongju-si, North Chungcheong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided